CLINICAL TRIAL: NCT02091284
Title: Prefrontal Modulation by Repetitive Bilateral Transcranial Direct Current Stimulation (tDCS) in Alcoholic Inpatients
Brief Title: Bilateral Prefrontal Modulation in Alcoholism
Acronym: tDCS_ALCOHOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Harvard Medical School (HMS and HSDM) (Other); University of Göttingen (Other)
Responsible Party: Principal Investigator, Ester Miyuki Nakamura-Palacios, MD, PhD, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS ALCOHOL CEP_UFES 384281; CNPq_ 475232/2013-5 (Other Grant/Funding Number: CNPq process # 475232/2013-5)
Record Dates: First submitted 2014-03-16; First posted 2014-03-19 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Drug Addiction; Executive Dysfunction
Keywords: alcoholism; tDCS; dlPFC; craving; cognition
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Sham-controlled double-blind randomized trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- real tDCS (Experimental): Ten sessions (every other day) of bilateral transcranial Direct Current Stimulation (tDCS: 2 milliamperes, 3 x 7 cm2, during 20 minutes) over dorsolateral Prefrontal Cortex (cathodal left / anodal right).
  Interventions: Device: transcranial Direct Current Stimulation
- sham-tDCS (Sham Comparator): Ten sessions (every other day) of placebo control (sham procedure) of transcranial Direct Current Stimulation (sham-tDCS) during 20 minutes with electrodes placed over the dorsolateral Prefrontal Cortex (cathodal left / anodal right). Current was delivered for 20 seconds and was turned off for the rest of the stimulation period. In this way, subjects experienced the initial itching sensation at the beginning of stimulation, but received no current for the rest of the session.
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — Direct currents were transferred via a pair of carbonated-silicone electrodes (35 cm2) with a thick layer of high conductive gel for EEG underneath them. The electric current will be delivered by an electric stimulator. To stimulate the left DLPFC, the cathode electrode was placed over F3 according to the 10-20 international system while the anode was placed over the contralateral F4 region. The currents flowed continuously for 20 minutes with an intensity of 2 milliamperes.
  Other Names: tDCS

SUMMARY:
In this study, eligible alcoholic inpatients recruited from a specialized clinic for addiction treatment, filling inclusion criteria and not showing any exclusion criteria, were randomized to receive the repetitive (10 sessions, every other day) bilateral dorsolateral Prefrontal Cortex (dlPFC: cathodal left / anodal right) tDCS (2 milliamperes, 5 x 7 cm2, for 20 min) or placebo (sham-tDCS). Craving to the use of alcohol was examined before (baseline), during and after the end of the tDCS treatment.

Based in our previous data, our hypothesis was that repetitive bilateral tDCS over dlPFC would favorably change craving in alcoholism and this would be a long-lasting effect.

DETAILED DESCRIPTION:
Before (baseline) and after tDCS or sham-tDCS treatment, subjects were clinically examined regarding craving (obsessive compulsive drinking scale) and they were followed-up for relapses at least 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients between the age of 18 and 60 years;
* met criteria for alcohol dependence according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV), as determined by clinical evaluation;
* in stable clinical condition with no need for inpatient care;
* able to read, write, and speak Portuguese; and
* no severe withdrawal signs or symptoms at baseline.

Exclusion Criteria:

* a condition of intoxication or withdrawal due to a substance other alcohol;
* unstable mental or medical disorder or substance abuse or addiction other than alcohol dependence, except nicotine and/or caffeine;
* a diagnosis of epilepsy, convulsions, or delirium tremens during abstinence from alcohol;
* a previous history of drug hypersensitivity or adverse reactions to diazepam or other benzodiazepines and haloperidol;
* any contraindication for electrical brain stimulation procedures such as electronic implants or metal implants;
* suspected pregnancy for female participants;
* any contraindication for magnetic resonance procedures such as electronic implants, metal implants, claustrophobia, or permanent make-up or tattoo received within the previous 3 months;
* the presence of vascular, traumatic, inflammatory, or tumor injuries detectable by CT examination.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ester MN Palacios, MD, PhD, Study Director — Federal University of Espírito Santo
Locations (1):
- Federal University of Espírito Santo, Vitória, ES - Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] da Silva MC, Conti CL, Klauss J, Alves LG, do Nascimento Cavalcante HM, Fregni F, Nitsche MA, Nakamura-Palacios EM. Behavioral effects of transcranial direct current stimulation (tDCS) induced dorsolateral prefrontal cortex plasticity in alcohol dependence. J Physiol Paris. 2013 Dec;107(6):493-502. doi: 10.1016/j.jphysparis.2013.07.003. Epub 2013 Jul 25. PMID 23891741
- [Background] Nakamura-Palacios EM, Souza RS, Zago-Gomes MP, de Melo AM, Braga FS, Kubo TT, Gasparetto EL. Gray matter volume in left rostral middle frontal and left cerebellar cortices predicts frontal executive performance in alcoholic subjects. Alcohol Clin Exp Res. 2014 Apr;38(4):1126-33. doi: 10.1111/acer.12308. Epub 2013 Nov 20. PMID 24256621
- [Background] Klauss J, Penido Pinheiro LC, Silva Merlo BL, de Almeida Correia Santos G, Fregni F, Nitsche MA, Miyuki Nakamura-Palacios E. A randomized controlled trial of targeted prefrontal cortex modulation with tDCS in patients with alcohol dependence. Int J Neuropsychopharmacol. 2014 Nov;17(11):1793-803. doi: 10.1017/S1461145714000984. Epub 2014 Jul 10. PMID 25008145
- [Result] Klauss J, Anders QS, Felippe LV, Nitsche MA, Nakamura-Palacios EM. Multiple Sessions of Transcranial Direct Current Stimulation (tDCS) Reduced Craving and Relapses for Alcohol Use: A Randomized Placebo-Controlled Trial in Alcohol Use Disorder. Front Pharmacol. 2018 Jul 3;9:716. doi: 10.3389/fphar.2018.00716. eCollection 2018. PMID 30018558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: AUD patients of both genders were successively recruited between June of 2015 and January of 2018 from three specialized clinics for drug dependence treatment, one public and two privates, from the State of Espírito Santo, Brazil.
Period: Overall Study
Arm/Group | Real tDCS | Sham-tDCS
Started | 26 (Two subjects from this group discontinued the protocol, data from one subject could not be included.) | 23 (One subject from this group discontinued the protocol)
Completed | 23 | 22
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — unreliable data | 1 | 0

BASELINE CHARACTERISTICS:
Population: Socio-demographic characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS | Sham-tDCS | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (12.0) | 43.5 (10.2) | 44.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 18 | 19 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 11 | 12 | 23
  Race: Brown | 8 | 6 | 14
  Race: Black | 4 | 4 | 8
Years of education [Count of Participants; unit: Participants]
  Up to 5 | 13 | 9 | 22
  Between 6 to 9 | 1 | 4 | 5
  Between 10 to 13 | 5 | 5 | 10
  Above 13 | 3 | 4 | 7
  Not reported | 1 | 0 | 1
Employment situation [Count of Participants; unit: Participants]
  Formal job | 2 | 6 | 8
  Informal job | 2 | 0 | 2
  Unemployed | 11 | 10 | 21
  Freelance | 2 | 2 | 4
  Disease benefit | 3 | 0 | 3
  Not reported | 1 | 2 | 3
  Retired | 2 | 2 | 4
Marital state [Count of Participants; unit: Participants]
  Single | 15 | 7 | 22
  Married or common-law | 7 | 7 | 14
  Divorced | 0 | 6 | 6
  Widow | 1 | 1 | 2
  Not reported | 0 | 1 | 1
Tobacco use [Count of Participants; unit: Participants]
  Yes | 12 | 11 | 23
  No | 11 | 11 | 22
Age at onset of alcohol use [Mean (Standard Deviation); unit: years] | 15.5 (5.4) | 16.9 (6.0) | 16.2 (5.7)
Amount of alcohol used (drinks/day) [Mean (Standard Deviation); unit: drinks/day] | 20.3 (13.4) | 15.5 (15.0) | 17.9 (14.3)
Days of abstinence before study [Mean (Standard Deviation); unit: days] | 33.0 (12.4) | 32.9 (12.5) | 33.0 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Craving
Description: Five items from the original obsessive compulsive drinking scale, which are believed to reliably assess craving in a narrow sense were used. Questions of this brief scale allow quantification of thoughts and feelings (obsessions), and behavioral intentions, and are answered on a scale ranging from 0 to 4, resulting in a total score between 0 and 20. Higher scores reflect more severe craving. These items were applied at the beginning, during and at the end of the treatment with sham-tDCS or tDCS.
Time Frame: Five applications: first week before tDCS treatment (baseline), second, third and fourth weeks, during the treatment, and in the fifth week, after the end of the tDCS treatment.
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Real tDCS | Sham-tDCS
Number analyzed (Participants) | 23 | 22
scores
  Initial scores (1st week) | 5.522 (4.44) | 3.818 (4.468)
  During treatment (2nd week) | 4.391 (3.751) | 4.136 (4.549)
  During treatment (3rd week) | 3.348 (3.485) | 3.545 (3.961)
  During treatment (4th week) | 1.739 (2.544) | 3.273 (4.322)
  Final scores (5th week) | 1.565 (2.409) | 2.455 (3.674)
Statistical Analysis 1: Comparison: Real tDCS vs Sham-tDCS; Test type: Other; p < 0.01, ANOVA — Two-way ANOVA with repeated measures followed by Bonferroni's multiple comparisons as post-hoc test and linear regression analyses. Additional comparisons between initial and final OCDS scores were done by paired t tests for each group
Statistical Analysis 2: Comparison: Real tDCS vs Sham-tDCS; Additional comparisons between initial and final OCDS scores were done by paired t tests for each group, and differences between final and initial scores were compared between sham-tDCS and tDCS groups with unpaired t tests; Test type: Other; p < 0.05, t-test, 2 sided

2. Other Pre Specified Outcome: Changes in Frontal Assessment Battery (FAB) Scores
Description: The FAB was used to explore six different domains of executive function. Each of these items is scored from 0 (zero) to a maximum of 3. Thus, the maximum score, meaning better scores, of FAB is 18. A single well trained examiner administered this assessment.
Time Frame: Before tDCS treatment (initial) and after the end of the tDCS treatment (final)
Measure: Mean (Standard Deviation); unit: scores
Groups:
- Sham-tDCS: Ten sessions (every other day) of placebo control (sham procedure) of transcranial Direct Current Stimulation (sham-tDCS) during 20 minutes with electrodes placed over the dorsolateral Prefrontal Cortex (cathodal left / anodal right).
Arm/Group | Real tDCS | Sham-tDCS
Number analyzed (Participants) | 23 | 22
scores
  initial | 12.48 (4.19) | 11.14 (2.95)
  final | 13.26 (4.41) | 13.32 (3.59)

3. Other Pre Specified Outcome: Changes in Mini-Mental Status Examination (MMSE)
Description: An adapted version of the MMSE in Portuguese was used. This version included an 11-item examination that examined five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score, meaning better scores, that could be achieved was 30, while a mean score between 23 and 26 or between 26 and 29 would be expected according to the age and educational level of the alcoholics.
Time Frame: Before tDCS treatment (initial) and after the end of the tDCS treatment (final)
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Real tDCS | Sham-tDCS
Number analyzed (Participants) | 23 | 22
scores
  initial | 23.13 (8.67) | 24.91 (5.82)
  final | 23.87 (8.42) | 24.64 (5.9)

4. Other Pre Specified Outcome: Changes in Hamilton Depression Rating Scale (HAM-D)
Description: A structured multiple-choice questionnaire was used to assess the severity of depression symptoms. This instrument assesses the severity of symptoms observed in depression, such as low mood, insomnia, agitation, anxiety and weight loss (Hamilton, 1960). Each question has between 3 and 5 possible answers that increase in severity. In the original scale, the first 17 questions contribute to the total score, while questions 18 to 21 provide additional information about depression (e.g., diurnal variation, paranoid symptoms), but are not included in the total score of the scale. Scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score is 52.
Time Frame: Before tDCS treatment (initial) and after the end of the tDCS treatment (final)
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Real tDCS | Sham-tDCS
Number analyzed (Participants) | 23 | 22
scores
  initial | 2.95 (2.1) | 3.0 (1.75)
  final | 2.17 (1.88) | 2.73 (2.25)

5. Other Pre Specified Outcome: Changes in Hamilton Anxiety Rating Scale (HAM-A)
Description: A structured multiple-choice questionnaire designed to assess the severity of anxiety symptoms was employed. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (e.g., mental agitation and psychological distress) and somatic anxiety (e.g., physical complaints related to anxiety). The higher the scores, higher the severity. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where below 17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: Before tDCS treatment (initial) and after the end of the tDCS treatment (final)
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Real tDCS | Sham-tDCS
Number analyzed (Participants) | 23 | 22
scores
  initial | 4.26 (5.9) | 3.77 (3.93)
  final | 3.87 (7.51) | 3.91 (6.36)

6. Other Pre Specified Outcome: Changes in Event-Related Potentials (ERPs)
Description: Electrophysiological recording was obtained through a 32-channel system placed on the scalp according to the International 10/20 EEG system.
  A cue-reactivity paradigm was adapted following standard cue-reactivity paradigms well established for pictures and videos. During picture presentation the subjects were asked to press a button whenever the drug-related pictures were presented, and to withhold the response when the neutral pictures were presented (50% of the time). The percent change of ventral medial Prefrontal Cortex current density was analyzed.
Time Frame: Before tDCS treatment (initial) and after the end of the tDCS treatment (final)
Population: ERP data was not possible in the total sample of each group because of technical difficulties.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Real tDCS | Sham-tDCS
Number analyzed (Participants) | 10 | 8
percent change | -30.34 (28.68) | 125.7 (141.6)

7. Other Pre Specified Outcome: Changes in Quality of Life of the World Health Organization (WHOQOL-BREF)
Description: An abbreviated instrument of cross-culturally valid assessment of quality of life of the World Health Organization (WHOQOL-BREF) with 26 questions translated to Portuguese was applied at the beginning and at the end of the five-week treatment. This instrument yields four domains (physical health, psychological, social relationships and environment) and two individually scored items regarding overall perception of quality of life (Q1, i.e., first question) and health (Q2, i.e., second question). The four domain scores are scaled in a way that higher scores stand for higher quality of life. These scores were transformed to be comparable with the scores used in the WHOQOL-100.
Time Frame: Before tDCS treatment (initial) and after the end of the tDCS treatment (final)
Population: These data was not collected correctly.
Arm/Group | Real tDCS | Sham-tDCS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were examined once at the end of each tDCS application. Therefore, over 10 tDCS applications, with a total of 10 examinations.
Description: We asked subjects about the following adverse effects: headache, neck and scalp pain, tingling, itching, skin redness, burning sensation of the scalp, sleepiness, acute mood changes, trouble concentrating, and others after treatment.
Arm/Group | Real tDCS | Sham-tDCS
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 16/23 | 13/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real tDCS (N=23) | Sham-tDCS (N=22)
Tingling in the scalp (Skin and subcutaneous tissue disorders) | 16 (16) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT02091284/Prot_SAP_000.pdf